CLINICAL TRIAL: NCT04040127
Title: Effect of Residual Dental Pulp Tissue and Cord Blood Stem Cells on Regeneration of Dental
Brief Title: Residual Dental Pulp Tissue and Cord Blood Stem Cells
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not obtain IRB approval
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-27622
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpal regeneration; Stem cells; Residual Pulpal Tissue; Irreversible Pulpitis
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The experiments outlined in this proposal are designed to test the hypothesis that the in vivo injection of cord blood stem cells (InvitRx®) into the root canal system will facilitate teeth initially diagnosed with irreversible pulpitis, to form normal healthy pulpal tissue.
Who Masked: Participant, Care Provider
Masking Description: Syringe with the intervention and control will be covered with masking tape in order for both the provider and the participant to be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cord blood stem cells (Experimental): cord blood stem cells from Invitrx
  Interventions: Biological: Cord blood stem cells
- 0.9% sodium chloride (saline) (Placebo Comparator): canal will be rinsed by saline solution.
  Interventions: Other: Saline solution

INTERVENTIONS:
Biological: Cord blood stem cells — Umbilical cords are collected from eligible donors at the time of delivery and transported to the processing facility on ice (2-8℃) in Dulbecco's Modified Eagle Media (DMEM). Cords are processed immediately under aseptic conditions and MSCs are collected for culture. Culture is maintained this way until the target number of cells has been reached, at which point passaged cells are suspended in Stem Cellbanker (Amsbio, Cambridge, MA) and frozen at -80℃.
  Arms: Cord blood stem cells
Other: Saline solution — saline solution used to rinse the canal.
  Arms: 0.9% sodium chloride (saline)

SUMMARY:
The experiments outlined in this proposal are designed to test the hypothesis that the in vivo injection of cord blood stem cells (InvitRx®) into the root canal system will facilitate teeth initially diagnosed with irreversible pulpitis, to form normal healthy pulpal tissue.

DETAILED DESCRIPTION:
Patients will be recruited from the various dental clinics at UCSF (student clinic, Advanced Education in General Dentistry clinic, post-graduate endodontics clinic, etc) that meet the inclusion and exclusion criteria. Patients in the control group will have root canal therapy initiated; instrumentation and cleaning up to 4mm from the radiographic apex. Bleeding will be induced and blood clot formed 3mm from the CEJ. MTA followed by glass ionomer and composite will be placed over the clot. Patients in the experimental group will have root canal therapy initiatied; instrumentation and cleaning up to 4mm from the radiographic apex. Bleeding will be induced and blood clot formed 3mm from the CEJ. 1 cc (30 million cord blood stem cells) will then be injected into the clot formation. MTA followed by glass ionomer and composite will be placed over the clot.

ELIGIBILITY:
Inclusion Criteria:

A. Patients must be systemically healthy, Class I dental category. B. Involved teeth must have no periodontal disease detectible by periodontal examination.

C. Patients must present without radiographic signs of endodontic disease (i.e. no periapical radiolucencies).

Exclusion Criteria:

A. Presence of any disease or medication that alters the immune system or interferes with healing ability B. Smokers (more than 10 cigarettes per day) C. External or internal tooth resorption D. Tooth perforation from the pulp cavity through the tip of the root exposing the tissue to material in the oral cavity.

E. Pregnant or nursing mothers because hormonal factors may influence the condition.

F. Allergies or adverse reactions to local anesthetic medications G. Patients under the age of 18. H. Patients with an ASA Classification II or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Regeneration of pulp | 6-9 months
  Absence of clinical symptoms and signs as well as response to thermal testing.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sabeti, DDS, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No